CLINICAL TRIAL: NCT04265768
Title: Dimensional Soft Tissue Changes Around Dental Implants Following the Use of a Collagen Matrix or a Connective Tissue Graft. A Pilot Study
Brief Title: Soft Tissue Changes Around Dental Implants
Acronym: Geistlich
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen Mary University of London (Other)
Collaborators: Geistlich Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRAS 268553
Record Dates: First submitted 2020-01-23; First posted 2020-02-12 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Tooth Loss; Dental Diseases; Wound Heal
Keywords: soft tissue regeneration; soft tissue graft; dental implant; imaging
MeSH Terms: conditions — Tooth Loss; Stomatognathic Diseases

STUDY DESIGN:
Intervention Model Description: The study will includes 3 groups randomised in parallel.
Who Masked: Outcomes Assessor
Masking Description: Due to the nature of the intervention, both participants and clinicians performing the surgical intervention will be un-blinded.
  Conversely, outcome examiners will be blinded to treatment allocation throughout the whole study duration.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- No Soft tissue augmentation surgery (Placebo Comparator): No soft tissue augmentation concomitant to implant placement. Negative control group.
  Interventions: Procedure: No soft tissue augmentation
- Soft tissue augmentation surgery with Fibro-Gide (Experimental): Soft tissue augmentation concomitant to implant placement with a porcine, volume-stable cross-linked collagen matrix (Fibro-Gide, Geistlich Pharma AG, Wolhusen, Switzerland).
  Test group.
  Interventions: Procedure: Soft tissue augmentation surgery with Fibro-Gide
- Soft tissue augmentation surgery with patient's CTG (Active Comparator): Soft tissue augmentation concomitant to implant placement with a connective tissue graft (CTG) taken from the patient's palate or retromolar area.
  Positive control group.
  Interventions: Procedure: Soft tissue augmentation surgery with CTG

INTERVENTIONS:
Procedure: Soft tissue augmentation surgery with CTG — An epithelial-connective tissue graft of approximately 2-3 mm of thickness and adequate length will be taken from the palate or retromolar region of the patient and de-epithelialized with a scalpel (ideally a thickness of 1.5-2.0mm).
  The connective tissue graft (CTG) obtained will then be positioned buccally to the dental implant and sutured to the internal side of the flap so to provide soft tissue bulk at the level of the neck of the implant and simulate a root prominence for the missing tooth.
  Arms: Soft tissue augmentation surgery with patient's CTG
Procedure: Soft tissue augmentation surgery with Fibro-Gide — Fibro-Gide will be used to obtain buccal soft tissue augmentation. Fibro-Gide will be trimmed with a scalpel and adjusted in size and thickness to better adapt to the area buccal to the implant. In particular, the graft will be shaped in order to obtain a graft of approximately 2-3 mm of thickness and adequate length. Fibro-Gide will then be sutured to the inner side of the buccal flap, before repositioning the flap and suturing it in a tension-free way.
  Arms: Soft tissue augmentation surgery with Fibro-Gide
Procedure: No soft tissue augmentation — During implant placement surgery, no soft tissue augmentation will be performed
  Arms: No Soft tissue augmentation surgery

SUMMARY:
This study aims to characterize the healing pattern following soft tissue augmentation procedure concomitant to implant placement.

DETAILED DESCRIPTION:
This study will characterize, for the first time, the healing pattern of soft tissues around dental implants in case of soft tissue augmentation and in comparison, to normal healing.

An innovative and comprehensive geometric/thermal imaging analysis will be employed that is non-contact and non-invasive to patients and will allow to characterize the healing process in a 2D-3D dimensional and volumetric way.

This approach, combined with LSCI and clinical and radiographic outcomes, will provide new data on the biology and critical phases of soft tissue healing around implants, as well as on the stability and aesthetics of the peri-implant tissues with different grafts.

Patient-reported outcome measurements (PROMs) will also be used to assess the level of pain and discomfort associated with soft tissue augmentation procedures.

ELIGIBILITY:
Inclusion Criteria:

* Age between 20 and 80 years.
* Good medical and psychological health.
* Absence of untreated caries lesions and untreated/uncontrolled periodontal disease. If patients require periodontal treatment (non-surgical and/or surgical), this has to be arranged outside the study protocol and completed at least 30 days prior to the enrolment.
* Need of a single-tooth replacement in the aesthetic (incisor, canine or premolar) region.
* Presence of adequate bone for implant placement without need for significant bone regeneration. In particular, the patients should have a bucco-palatal residual alveolar width of at least 6 mm at the central and crestal aspect of the single tooth gap to ensure complete embedding of an implant by bone (De Bruyckere et al., 2018).
* A residual alveolar height >8 mm, enough inter-arch space for a crown and a minimum distance of 6 mm from the adjacent teeth.
* The width and height will be confirmed after x-ray examination in Visit 1 (or extra visit). Cases of small apical fenestration (≤ 25% of implant length) after implant placement will not be excluded, but will be treated according to the GBR principle (collagen membrane associated with a deproteinized bovine bone graft) to re-establish the bone contour and without over contouring.
* At least 8 weeks of post-extraction socket healing had occurred in the edentulous site.
* Willingness to sign the informed consent form.

Exclusion Criteria:

* Self-reported pregnancy and lactation.
* Any known systemic disease affecting bone metabolism (e.g. Cushing's syndrome, crohn's disease, rheumatoid arthritis, osteoporosis, diabetes type I and uncontrolled diabetes type II), systemic infections or recent surgical procedures within 30 days of study initiation.
* Chronic treatment (i.e., 2 weeks or more) with any medication known to affect oral status (e.g., phenytoin, dihydropyridine, calcium antagonists and cyclosporine) or bone metabolism (e.g. bisphosphonates, hormone replacement therapy, immunosuppressants) within 1 month before baseline visit.
* HIV or viral hepatitis.
* Physical handicaps that would interfere with the ability to perform adequate oral hygiene.
* Self-reported alcoholism or chronic drug abuse.
* Heavy smokers (>10/cigarettes per day).
* Patients suffering from a known psychological disorder or with limited mental capacity or language skills such that study information could not be understood, informed consent could be obtained or simple instructions could be followed.
* Full-mouth bleeding (BOP) and plaque (PI) scores >30% or sites with periodontal pocket depth >5 mm at the completion of the pre-treatment phase.
* Very thin or very thick biotypes that according to the clinician's judgement would either risk to have complications or would not benefit from receiving a graft.
* <2 mm KT buccally (from the mucogingival junction to the coronal aspect of the crestal soft tissue).

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2021-06-21 (Actual); Primary Completion 2025-02-24 (Actual); Study Completion 2025-02-24 (Actual)

PRIMARY OUTCOMES:
3D intra-oral volume changes in mucosal soft tissue following augmentation | Immediately after implant placement.
  Those changes will be assessed by capturing 3D intra-oral scans at the different time-points.
3D intra-oral volume changes in mucosal soft tissue following augmentation | 7, 14 and 30 Days post implant placement
  Those changes will be assessed by capturing 3D intra-oral scans at the different time-points.
3D intra-oral volume changes in mucosal soft tissue following augmentation | 12 weeks and 16 weeks post- implant loading.
  Those changes will be assessed by capturing 3D intra-oral scans at the different time-points.
3D intra-oral volume changes in mucosal soft tissue following augmentation | 12 month post- implant loading.
  Those changes will be assessed by capturing 3D intra-oral scans at the different time-points.

SECONDARY OUTCOMES:
Changes in gingival thickness | implant placement to 12 weeks after implant placement
  Changes in gingival thickness from the time of implant placement (with or without graft) and 12 weeks after implant placement assessed by a caliper
3D extra-oral volumetric changes | baseline, immediately after implant placement, 7, 14 and 30 days after implant placement
  3D extra-oral morphometric changes assessed with a facial scanner
2D-3D intra-oral thermal changes | baseline to 1, 3, 7, 14 and 30 days after implant placement
  2D-3D intra-oral thermal changes using an infrared, contact-free, thermal camera
changes in vascularisation | before and immediately after implant placement, and at post-operative days 1, 3, 7, 14, and 30
  Changes in revascularization in the area of the implant surgery with laser speckle contrast imaging
soft tissue aesthetics | At implant loading and at 12 months after loading.
  Papilla Fill Index and Pink Aesthetic Score
changes in height of keratinised tissue | baseline to 30 days, 12 weeks and 16 weeks after implant placement and 12 months post loading
  changes in height of keratinised tissue measured with a probe
Patients' reported outcomes (PROMS) in oral impact on Daily Performances (OIDP) questionnaire (OIDP) | At basline, 3 months (visit2, 3 and 4), 1 week from visit 2, 2 weeks form visit 2, 1 month from visit 2.
  The OIPD is a well validated and frequently used PROMs in studies of oral health. It is a composite measure of the impacts of oral health on the quality of life of people. The OIDP focuses on the impact of oral health on the quality of life of people. The OIDP focuses on the impact that the conditions of the teeth and social wellbeing of the person. More specifically, it assesses the impact of oral conditions on basic daily life activities and behaviours (eating, speaking, cleaning teeth, going out, relaxing, smiling, major work or role, emotional stability, social contact). For each performance, both the frequency and severity of oral impacts are assessed. The overall OIDP score ranges from 0 to 100, with higher scores indicating worse quality of life.
PROMs based on the evaluation of global changes in quality of life | At basline, 3 months (visit2, 3 and 4), 1 week from visit 2, 2 weeks form visit 2, 1 month from visit 2.
  Global ratings on health and quality of life will be provided through two methods:
  1. The Visual Analogue Scale (VAS) included in the EQ5D questionnaire.
  2. Through the following question: 'how would you rate the quality of your life'?
  The response will be scored on a six-point scale as:
  1. Excellent
  2. Very good
  3. Good
  4. Fair
  5. Poor
  6. Very poor
PROMs based on the evaluation of patient's perception about therapy | At basline, 3 months (visit2, 3 and 4), 1 week from visit 2, 2 weeks form visit 2, 1 month from visit 2.
  The extent of discomfort and/or pain experienced will be evaluated using a 100-mm horizontal visual analogue scale (VAS). The anchors for each end of the scales will be designated as none and extreme. Patients will be also instructed to quantify the analgesic medication taken. In addition, the extent of discomfort, root hypersensitivity, oedema, hematoma, high fever and interference in daily activities during the first post-therapy week will be evaluated in the same way.
Post-operative swelling and oedema | At basline, 3 months (visit2, 3 and 4), 1 week from visit 2, 2 weeks form visit 2, 1 month from visit 2.
  A series of subtracted images from the baseline will accurately identify the area and magnitude of the swelling, changes in facial shape, volume and temperature to monitor/quantify the healing. For every patient, a person specific template of postoperative facial swelling/oedema pattern will be created for sequential swelling/thermal changes or oedema volume measurements that will be applied on a unique alignment of the patient's specific consecutive imaging surfaces (self-defined positioning based on patients facial features).

CONTACTS AND LOCATIONS:
Overall Officials: Nikos Donos, PhD, Principal Investigator — Barts & The London School of Medicine & Dentistry, QMUL
Locations (2):
- United Kingdom (2):
  - Barts and The London Dental Hospital, London
  - Centre for Oral Clinical Research (COCR), London

IPD SHARING:
Plan to Share IPD: No